CLINICAL TRIAL: NCT01221883
Title: Early Pharmacological Intervention With Diazepam in the Emergency Room Setting to Prevent Posttraumatic Stress Disorder (PTSD).
Brief Title: Prevention of Posttraumatic Stress Disorder (PTSD) With Diazepam
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Pablo Roitman, MD, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ER DIAZEPAM PTSD- HMO-CTIL
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress; Prevention; Diazepam
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Diazepam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule in ER, identical follow up like those in the active arm.
  Interventions: Drug: Diazepam
- Diazepam (Experimental): 10 mg of Diazepam mg orally at ER only (a single administration)
  Interventions: Drug: Diazepam

INTERVENTIONS:
Drug: Diazepam — Single dose 10mg Diazepam tablet

SUMMARY:
PTSD is a pervasive and frequent disorder. Early psychological treatment - but not pharmacology - effectively prevent PTSD.

Current pharmacological studies did not include treatment given immediately after trauma exposure.

However, a recent study of opiates suggests that their early administration may reduce the likelihood of developing PTSD - possibly by mitigating early post-traumatic distress (UCR) - within an adequate window of time.

Benzodiazepines are often used to reduce anxiety and agitation during stressful situations - including traumatic event.

These compounds may increase the likelihood of developing PTSD when administered few days after the traumatic event - but their effect as an immediate intervention has not been studied - despite their frequent and uninformed use at this stage.

This work will evaluate the effect of diazepam - a BZ compound - on PTSD symptom trajectory following traumatic event in a randomized controlled design.

Following the studies of opiates it is hoped that diazepam, administered within hours of the traumatic event, and before the first night sleep (a memory consolidating condition) will reduce the likelihood of developing PTSD. However, an adverse effect cannot be excluded, and thus the investigators posit a bidirectional hypothesis.

The importance of this work is that it will provide the necessary evidence to sanction a frequently practiced use of benzodiazepines.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients that have experienced an acute event that meets the DSM-IV A.1 PTSD criterion: "the person experienced, witnessed, or was confronted with an event or events that involved actual or threatened death or serious injury, or a threat to the physical integrity of self or others;"
* Outpatients that also meet DSM-IV A.2. PTSD criterion: "the person's response involved intense fear, helplessness, or horror;" and
* Outpatients that have a heart rate upon ED presentation >80 BPM
* Outpatients that hadn't fallen asleep for a night after traumatic event before ED arrival;

Exclusion Criteria:

* Physical injury that requires hospitalization, interferes with a patient's ability to cooperate with screening or give informed consent, or otherwise contraindicates participation;
* Traumatic event reflecting ongoing victimization (e.g., domestic violence) to which the patient is likely to be re-exposed during the study period;
* Head injury with loss of consciousness or amnesia;
* Medical condition that contraindicates the administration of diazepam :

  * hepatic insufficiency, severe
  * hypersensitivity to diazepam
  * myasthenia gravis
  * narrow-angle glaucoma, acute
  * respiratory insufficiency, severe
  * sleep apnea syndrome
* Current use of medication that may involve potentially dangerous interactions with diazepam, including opioids, barbitals and another benzodiazepines; when used in combination, these drugs have additive CNS and respiratory depressant effects
* Women who are currently pregnant or nursing.
* Those at immediate risk of harming self or others; those who have a clinically significant medical illness or other significant psychiatric illness;
* Overt psychopathology, substance abuse/dependence, intoxication, odor of alcohol, or discernible substance effect;

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered Posttraumatic Scale (CAPS) | 20 minutes
  Is a structured clinical interview that evaluates the 17 DSM-IV PTSD and associated symptoms on dimensions of frequency and intensity (0-4 scale for each). The CAPS also includes measures of global response validity, global PTSD symptom severity, and impact of symptoms on occupational and global functioning. The CAPS contains explicit, behaviorally anchored prompt questions and rating scale descriptors to enhance reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organitation, Jerusalem, Israel

REFERENCES:
- [Background] Gelpin E, Bonne O, Peri T, Brandes D, Shalev AY. Treatment of recent trauma survivors with benzodiazepines: a prospective study. J Clin Psychiatry. 1996 Sep;57(9):390-4. PMID 9746445
- [Background] Meares S, Shores EA, Batchelor J, Baguley IJ, Chapman J, Gurka J, Marosszeky JE. The relationship of psychological and cognitive factors and opioids in the development of the postconcussion syndrome in general trauma patients with mild traumatic brain injury. J Int Neuropsychol Soc. 2006 Nov;12(6):792-801. doi: 10.1017/S1355617706060978. PMID 17064443